CLINICAL TRIAL: NCT00496574
Title: Evaluation of Long-term Clinical Efficacy of House Dust Mite Immunotherapy in Children With Bronchial Asthma
Brief Title: Evaluation of Efficacy of House Dust Mite Immunotherapy in Children With Bronchial Asthma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Iwona Stelmach, MD, PhD, Professor, Medical University of Lodz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RNN-102-06-KE
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Asthma
Keywords: asthma; immunotherapy; efficacy; children; symptoms score; quality of life; spirometry; PC20M
MeSH Terms: conditions — Asthma | interventions — Novo-Helisen Depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Biological: Novo Helisen Depot, Phostal
- 2 (No Intervention): no intevention

INTERVENTIONS:
Biological: Novo Helisen Depot, Phostal — subcutaneous immunotherapy
  Other Names: Novo Helisen Depot
  Arms: 1

SUMMARY:
The aim of the study is to assess the effect of specific immunotherapy (SIT) to dust mites on clinical symptoms, reliever drugs usage, inhaled glucocorticosteroid usage, quality of life, lung function, bronchial hyperreactivity with methacholine, and presence and type of allergy after three years of SIT in children with asthma.

DETAILED DESCRIPTION:
According to Global Initiative for Asthma treatment of asthma is based on avoidance of allergens, pharmacological treatment, and specific immunotherapy.

The aim of the study is to assess the effect of specific immunotherapy (SIT) to dust mites on clinical symptoms, reliever drugs usage, inhaled glucocorticosteroid usage, quality of life, lung function, bronchial hyperreactivity with methacholine, and presence and type of allergy after three years of SIT in children with asthma.

ELIGIBILITY:
Inclusion Criteria:

* patients allergic to house dust mites
* patients with moderate bronchial asthma
* patients with controlled asthma
* patients who were qualified for immunotherapy and gave written informed consent for immunotherapy (active treatment group)
* patients who were qualified for immunotherapy and did not agree with this kind of treatment - did not give written informed consent for immunotherapy (control group)

Exclusion Criteria:

* patients allergic for other perennial and seasonal allergens
* patients with other chronic diseases that either put the patient at risk when participating in the study or could influence the results of the study or the patient's ability to participate in the study as judged by the investigator
* medications that resulted in patient exclusion included:anti-parasites or oral corticosteroids within 6 months before the first visit.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-05; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
clinical symptoms, reliever drugs usage, inhaled glucocorticosteroid usage, quality of life, lung function | baseline (first visit), 12 months (second visit), 24 months (third visit), 36 months (fourth visit)

SECONDARY OUTCOMES:
bronchial hyperreactivity with methacholine, and presence and type of allergy after tree years of SIT in children with asthma. | after 36 months (fourth visit)

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Sobocińska, MD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, Lodz, Poland; Iwona Stelmach, MD PhD Prof, Study Chair — Department of Pediatrics and Allergy, Medical University of Lodz, Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz, Poland, Lodz, Poland